CLINICAL TRIAL: NCT06533462
Title: Infant Food Allergen Oral Immunotherapy (InFO)
Brief Title: Randomized Controlled Trial of Slow Multiallergen Oral Immunotherapy in Young Children
Acronym: InFO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Idun Holmdahl, Pediatrician, Postdoctoral researcher, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dnr 2024-03574-02
Record Dates: First submitted 2024-07-12; First posted 2024-08-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Food Allergy; Oral Immunotherapy for Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is blinded and neither participants nor the study team physicians know who is receiving multiallergen powder or placebo. Only few persons outside the study has this knowledge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Allergic children - Multiallergen OIT (Active Comparator): Children with food allergy receiving multiallergen powder OIT. Multiallergen food challenge is done before randomization and one and two years after inclusion. OIT multiallergen powder with slow up-dosing until 3 teaspoons of the multiallergen powder is reached and taken daily. 2 years treatment.
  Number = 40 patients
  Intervention: multiallergen powder
  Interventions: Dietary Supplement: Multiallergen powder
- Group B: Allergic children - Placebo powder (No Intervention): Children with food allergy receiving OIT with placebo powder (gluten-free oatmeal). Multiallergen food challenge is done before randomization and one and two years after inclusion.
  Number = 40 patients
- Group C: Non-allergic children - low dose multiallergen powder (Active Comparator): Children not reacting to the baseline challenge who will be randomized to eat a low dose of the multiallergen powder, 1 teaspoon daily. Multiallergen food challenge is done before randomization and one year after inclusion. 1 year treatment.
  Number = X
  Intervention: Multiallergen powder
  Interventions: Dietary Supplement: Multiallergen powder
- Group D: Non-allergic children - placebo powder (No Intervention): Children not reacting to the baseline challenge who will be randomized to eat placebo powder (gluten-free oatmeal) and no specific advice.
  Number= X

INTERVENTIONS:
Dietary Supplement: Multiallergen powder — OIT multiallergen powder.
  Arms: Group A: Allergic children - Multiallergen OIT; Group C: Non-allergic children - low dose multiallergen powder

SUMMARY:
The aim is to study whether a multiallergen oral immunotherapy (OIT) strategy with slow up-dosing and low treatment dose against food allergy in young children (0.5-3 years) is safe and effective, a method to cure food allergy and to prevent the development of new food allergies.

Clinical randomized controlled (1:1) blinded interventional trial (RCT) with 2 intervention arms (group A and B).

Among 80 children reacting at the multiallergen food challenge, 40 children will be randomized to receive OIT (oral immunotherapy) with multiallergen powder with a final dose of approximately 200 mg protein of each included food (egg, milk, soy, wheat, walnut, peanut, hazelnut, cashew, almond, lentils)(group A) or to receive placebo powder (gluten-free oatmeal) (group B).

A sub-analysis will be performed of the children not reacting to the baseline challenge, who will be randomized to eat a low dose of the multiallergen powder (group C) or placebo powder (gluten-free oatmeal) (group D) and no specific advice.

DETAILED DESCRIPTION:
Today, there is no established curative treatment for food allergies, and those affected must avoid the food that triggers symptoms. The most studied method is oral immunotherapy (OIT) which have mainly been carried out on children >4 years of age. The OIT method implies that the allergic individual eats initially very low doses and gradually increasing amounts of the allergen until a maintenance dose is reached. The treatment aims to induce desensitization or tolerance to the allergen.

Intervention: The intervention substance is a powder containing a prespecified amount of 10 allergens (egg, milk, wheat, lentils, soy, walnut, peanut, hazelnut, cashew, almond), which are the most triggering allergens in children. The product is developed in cooperation with Research Institute of Sweden (RISE).

Clinical randomized controlled (1:1) blinded interventional trial (RCT) with 2 interventions arms (group A and B). A sub-analysis will be performed of the children not reacting to the baseline challenge (group C and D).

Group A: Children with food allergy (sensitization and positive baseline challenge), receiving multiallergen powder OIT, slow up-dosing until 3 teaspoons of the multiallergen powder is reached daily. Food challenge will be performed after 1 and 2 years. 2 years treatment.

Group B: Children with food allergy (sensitization and positive baseline challenge), receiving OIT with placebo (gluten-free oatmeal) followed by maintenance, in total 2 years. Food challenge will be performed after 1 and 2 years.

Group C and D: sensitized children with a negative baseline challenge will be randomized 1:1 for treatment with multiallergen powder or placebo powder in a lower amount, 1 teaspoon daily and can introduce food in accordance with Swedish guidelines. After one year a food challenge will be performed.

Selection for group A to D: All children 0.5-3 years of age in Stockholm County who had a positive blood test for suspected food allergy to one or more of the 10 included allergens with specific immunoglobulin E (IgE) >0.1 kUA/L, are eligible as possible study participants. The data is obtained from the Karolinska University Laboratory's test results register. Information letters will be sent to families with IgE-sensitized children.

Inclusion groups A to D: Children 0.5-3 years old at inclusion with positive IgE >0.1 kUA/L against at least one of the 10 above mentioned allergens. Eighty children, group A (n=40) and group B (n=40) also need a positive baseline food challenge.

Children with a negative food challenge (group C and D) (number is not determined) do not react at the baseline challenge.

Primary outcome: Tolerance to 900 mg protein, cumulative dose, of each of the 10 included allergens, at the food challenge after two years OIT treatment or placebo (group A and B).

Secondary outcomes: Tolerance to cumulative dose of 900 mg protein of each food, evaluated with a food challenge after one years in all children (group A-D). Changes in immunological markers, eczema and asthma status and changes in quality of life in relation to interventions.

ELIGIBILITY:
Inclusion Criteria:

* 0.5-3 years old at inclusion with IgE (>0.1 kUA/l) against at least one allergen (wheat, lentils, egg, milk, soy, walnut, hazelnut, peanut, almond, cashew).
* Written consent for participation in the study for both guardians.
* 80 children (group A and B) also need a positive baseline food challenge.
* Children with a negative food challenge (group C and D) (number not determined) do not react at the baseline challenge.

Exclusion Criteria:

* other serious illness
* previous life-threatening anaphylaxis (intensive care)
* eosinophilic esophagitis
* eosinophilic gastrointestinal disease
* severe chronic gastroesophageal reflux disease
* unclear recurrent GI complaints
* low body weight <2SD
* participation in another intervention study if included in intervention group
* severe uncontrolled asthma
* medication with biological drugs or oral steroids.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Tolerance to 900 mg protein at a food challenge after 2 years | 2 years
  Tolerance to 900 mg protein, cumulative dose, of each of the 10 included allergens (in the multiallergen powder), evaluated at a food challenge after 2 years in group A and B. Tolerance is defined as no objective sign of an allergic symptom (urticaria, flush, swelling/angioedema, nasal symptoms, eye symptoms, hoarseness, muffled speech, persistent cough, wheezing, stridor, persistent abdominal pain, severe nausea, vomiting, diarrhea, general impact, drop in blood pressure, decreased oxygenation saturation) within 2 hours after the last dose during the food challenge after 2 years of OIT/placebo.

SECONDARY OUTCOMES:
Tolerance to cumulative dose of 900 mg protein at a food challenge after 1 year | 1 year
  Tolerance to cumulative dose of 900 mg protein of each of the 10 included allergens in the multiallergen powder, evaluated at a food challenge after one year in all children (A, B, C, D).
  Tolerance is defined as no objective sign of an allergic symptom (urticaria, flush, swelling/angioedema, nasal symptoms, eye symptoms, hoarseness, muffled speech, persistent cough, wheezing, stridor, persistent abdominal pain, severe nausea, vomiting, diarrhea, general impact, drop in blood pressure, decreased oxygenation saturation) within 2 hours after the last dose during the food challenge after one year.
Oral brush samples | 1 and 2 years
  The oral microbiome will be investigated with sequencing-based methods to monitor possible changes in the oral microbiota composition and function related to OIT treatment. Comparisons will be made between intervention groups and analyzed in relation to intervention. Oral brush samples will be collected in connection with the visit for the baseline challenge, at the challenge at 1 years (group A-D) and 2 years (group A-B).
Intestinal microbiome | 1 and 2 years
  The gut microbiome will be investigated with sequencing-based methods to monitor possible changes in the gut microbiota composition and function related to OIT treatment. Comparisons will be made between intervention groups and analyzed in relation to intervention. Fecal samples will be collected in connection with the visit for the baseline challenge, at the challenge at 1 years (group A-D) and 2 years (group A-B).
Immunological biomarkers | 1 and 2 years
  To study different immunological biomarkers (e.g. T-helper cell population and polarization and IgE-levels) before, during and after OIT treatment and compare this to the placebo group. Immunological marker in mononuclear cells in peripheral blood will be analyzed ex vivo with flowcytometri and RNA-sequencing platforms. Circulating immunological factors, e.g. cytokines and chemokines will be analyzed in plasma with ELISA-based methods. Mononuclear cellpopulations in peripheral blood will be exposed to different stimuli (such as sensitizing allergen, anti-C D3/ C D28) in vitro, type and level of reaction in the different cellpopulations will be monitored at mRNA- and protein-level.
  Blood sampling will be collected in connection with the visit for the baseline challenge, at the challenge at 1 years (group A-D) and 2 years (A-B).
Changes in eczema status in relation to interventions | 1 and 2 years
  Clinical examination including eczema grading will be performed at the food challenges and basic clinical examination at each study-visit. Eczema grading will be evaluated using Eczema area and severity index (EASI), score between 0-72.
Changes in asthma status in relation to interventions | 1 and 2 years
  Clinical examination including evaluation asthma status will be performed at the food challenges and basic clinical examination at each study-visit. Asthma status will be evaluated with a clinical examination, use of asthma medication, number of wheezing episodes as well as hospitalization prior to the study visit.
Changes in quality of life in relation to interventions | 1 and 2 years
  To evaluate changes in quality of life before and after multiallergen OIT using the "Food allergy quality of life questionnaire-parental form" (FAQLQ-PF) validated and translated into Swedish. Comparisons will be made between the OIT group and the placebo group. FAQLQ-PF is a multidimensional parent report measure to assess children between 0-12 years. There are 14 items for children below 4 years old which are scored on a 7 point scale from 0 (no impact of HRQL) to 6 (extreme impact of HRQL). FAQLQ-PF include questions for food-allergy specific QoL with general emotional impact, food anxiety, social and dietary limitations. Overall and domain specific HRQL scores will be calculated. Higher score mean worse outcome and a score of ≥ ±0.5 will be considered clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nilsson, MD, PhD, Principal Investigator — Karolinska Institutet; Anna Asarnoj, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No